CLINICAL TRIAL: NCT00992043
Title: Efficacy and Safety of Creatine Supplementation Combined With Exercise Training in Type 2 Diabetic Patients
Brief Title: Creatine Supplementation and Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Bruno Gualano, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: eefeusp2
Record Dates: First submitted 2009-10-07; First posted 2009-10-08 (Estimated); Last update posted 2010-03-23 (Estimated); Status verified 2009-10

CONDITIONS: Diabetes; Renal Function
Keywords: creatine supplementation; exercise training
MeSH Terms: conditions — Diabetes Mellitus | interventions — Creatine; Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- exercise and placebo (Placebo Comparator)
  Interventions: Dietary Supplement: creatine; Other: Exercise training
- exercise and creatine (Experimental)
  Interventions: Dietary Supplement: creatine; Other: Exercise training

INTERVENTIONS:
Dietary Supplement: creatine
Other: Exercise training

SUMMARY:
Creatine supplementation is capable of improving glucose tolerance in healthy subjects. The researchers aim to investigate whether this supplement can affect metabolic control in diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* males and females type 2 diabetic patients
* glycated hemoglobin between > 9%
* non insulin users
* physically inactive
* only metformin and/or sulfonylurea users
* BMI > 30 kg/m2
* age of years > 50 y

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2009-10; Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
glycated hemoglobin | three months

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Gualano, PhD ongoing, Principal Investigator — University of Sao Paulo
Locations (1):
- General Hospital - School of Medicine - University of Sao Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Gualano B, Lugaresi R, de Salles Painelli V, Queiroz AC, Artioli G, Roschel H, Otaduy MC, Leite Cda C, Lancha AH Jr. Creatine supplementation does not augment muscle carnosine content in type 2 diabetic patients. Appl Physiol Nutr Metab. 2011 Oct;36(5):764-7. doi: 10.1139/h11-083. PMID 21999299
- [Derived] Gualano B, de Salles Painelli V, Roschel H, Lugaresi R, Dorea E, Artioli GG, Lima FR, da Silva ME, Cunha MR, Seguro AC, Shimizu MH, Otaduy MC, Sapienza MT, da Costa Leite C, Bonfa E, Lancha Junior AH. Creatine supplementation does not impair kidney function in type 2 diabetic patients: a randomized, double-blind, placebo-controlled, clinical trial. Eur J Appl Physiol. 2011 May;111(5):749-56. doi: 10.1007/s00421-010-1676-3. Epub 2010 Oct 26. PMID 20976468